CLINICAL TRIAL: NCT03536715
Title: Qualitative Patient Interviews to Develop a Patient-Reported Outcomes (PRO) Instrument to Assess Visual Symptoms in KAMRA® Inlay Patients
Brief Title: Qualitative Validation of Patient-Reported Outcomes (PRO) Instrument
Status: Completed | Type: Observational
Sponsor: AcuFocus, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: KAMR-201-PRO1
Record Dates: First submitted 2017-11-09; First posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Patient-Reported Outcomes (PRO)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to conduct concept elicitation and cognitive debriefing interviews with patients who have been implanted with the KAMRA inlay in order to assess the content validity of a PRO instrument

ELIGIBILITY:
Inclusion Criteria:

1. Minimum 45 years of age, maximum age 60 years;
2. Subject has been implanted with the KAMRA inlay;
3. Subject is in good general health, as evidenced by medical history;
4. Subject is willing and able to attend and participate in the interviews and demographic questionnaire (fluent in U.S. English); and
5. Signed informed consent document.

Exclusion Criteria:

1. Subject has severe neurological or cognitive deficits or an uncontrolled psychiatric condition that might affect their ability to participate in the interview;
2. Subject has insufficient ability to read or write that would prevent them from completing a questionnaire without help;
3. Subject is not a fluent speaker of U.S. English; or
4. Subject is unable to attend the interview.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The sample recruited will reflect the target KAMRA inlay patient population. Thus, a minimum of 20 subjects (up to 50 subjects to achieve saturation) who have been implanted with the KAMRA inlay will be recruited from up to 5 sites across the US. Subjects with a range of post-operative experience, satisfaction, visual symptoms, ages and educational abilities will be recruited. In addition, subjects who are of non Caucasian ethnicity will be included.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

PRIMARY OUTCOMES:
PRO instrument | 6 months
  Develop PRO instrument that will assess KAMRA inlay-related visual symptoms and to establish the content validity of that PRO instrument.